CLINICAL TRIAL: NCT05517863
Title: The Effect of Combined 650 nm and Infrared Laser on Chronic Diabetic Foot Ulcer Surface Area: a Randomized Controlled Trial
Brief Title: The Effect of Combined 650 nm and Infrared Laser on Chronic Diabetic Foot Ulcer Surface Area:
Acronym: wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidy F. Ahmed (Other)
Responsible Party: Sponsor-Investigator, Heidy F. Ahmed, Doctor of physical therapy at Al kasr Al Anini teaching hospital, Cairo, Egypt, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LASER.REC/2022
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Foot; Wound Heal
Keywords: 650 nm laser; infrared laser; chronic diabetic foot ulcer; wound surface area
MeSH Terms: conditions — Diabetic Foot | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive traditional wound care
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient didn't know the types of modes of laser applied even in the control group i used light not laser to equalize the blindness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laser sequential mode (Experimental): All patients received 2 sessions of laser therapy / week with different wavelengths in sequential mode in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care
  Interventions: Device: laser therapy
- laser seperate mode (Experimental): All patients received 2 sessions of laser therapy / week with different wavelengths in seperate mode in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care
  Interventions: Device: laser therapy
- traditional wound care (Active Comparator): (II) Traditional wound care inform of
  1. Wound care treatment
     * Debridement to remove necrotic tissue
     * Irrigation of the wound by normal saline
     * Change dressing daily to protect wound from infection
  2. Foot care
     * Wash feet daily, dry carefully especially between toe
     * Avoid extreme temperatures
     * Inspection daily of foot blisters
  3. Foot wear
     * Avoid walking bare foot
     * Properly fitted shoes
     * Avoid wearing open-toed shoes
  Interventions: Device: laser therapy

INTERVENTIONS:
Device: laser therapy — All patients received 2 sessions of laser therapy / week in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care:
  (I) Use red & infrared laser therapy device with 4 different wavelengths in a synchronized mode:
  1. 980 nm for wound decontamination, improve circulation, lymphatic drainage
  2. 915 nm enhances O2 delivery
  3. 810 nm increases ATP production
  4. 650 nm accelerate surface healing, tissue regeneration plus traditional wound treatment mentioned before

SUMMARY:
Objective: investigate the effect of combined 650 nm and infrared laser on chronic diabetic foot ulcer surface area.

Participants: The forty five patients will assigned randomly into three equal groups, each group consist of 15 patients, group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive traditional wound care

DETAILED DESCRIPTION:
Objective: investigate the effect of combined 650 nm and infrared laser on chronic diabetic foot ulcer surface area.

Participants: The forty five patients will assigned randomly into three equal groups, each group consist of 15 patients, group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive traditional wound care Outcomes: the primary outcomes were the wound surface area measurement, % of wound complete closure and % of days needed for surface area reduction before and after receiving the treatment protocol for two consequetive months, and the secondary outcomes were % of wound cause and location frequencies

ELIGIBILITY:
Inclusion Criteria:

* 1- Diabetic patients with either type I or II 2- Age from 18-60 years old, both sexes 3- Ulcer lasting longer than two months 4- DFU grade 1 or 2 according to Wagner classification. 5- All patients able to walk dependently

Exclusion Criteria:

1. Patients with vascular disease
2. Patients with fixed ankle deformity as Charcot foot or stiffness
3. Patients with any type of osteomyelitis associated with DFU
4. Patients with renal or hepatic failure
5. BMI < 30 kg/m2 as Obesity can cause poor perfusion due to vascular insufficiencies; altered population of immune mediators may lengthen the inflammatory process & decrease oxygenation of subcutaneous adipose tissue which is liable to be infected.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
percent of wound size measurement methods | two consecutive months
  weekly by
  1. a ruler (wound area was calculated by measuring and multiplying the greatest length by the greatest width perpendicular to the greatest length)
  2. a sterile transparent film sheet
percent of wounds complete closure | two consecutive months
  measure percent of wounds complete closure in each group

SECONDARY OUTCOMES:
percent of each type of wound cause | two consecutive months
  different wound cause diabetic foot ulcers and healing time
percent of each wound location | two consecutive months
  different wound location in diabetic foot ulcers and healing time
percent of days needed for surface area reduction | two consecutive months
  measure the days needed to decrease surface area in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S El Basiouny, Principal Investigator — national institute of laser sciences; Heidy F Ahmed, master, Principal Investigator — Kasr al aini
Locations (1):
- National Institute of Laser Sciences, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), all IPD that underline results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In the next month of registration.
Access Criteria: Information will be available upon request through the following e-mail: heidy.fouad@gmail.com.

REFERENCES:
- [Background] Experimental Study of the Effect of Photobiomodulation Therapy on the Regulation of the Healing Process of Chronic Wounds
- [Background] Hamblin, M. R., Agrawal, T., & de Sousa, M. (Eds.). (2016). Handbook of low-level laser therapy. CRC Press.
- [Background] Rupel K, Zupin L, Colliva A, Kamada A, Poropat A, Ottaviani G, Gobbo M, Fanfoni L, Gratton R, Santoro M, Di Lenarda R, Biasotto M, Zacchigna S. Photobiomodulation at Multiple Wavelengths Differentially Modulates Oxidative Stress In Vitro and In Vivo. Oxid Med Cell Longev. 2018 Nov 11;2018:6510159. doi: 10.1155/2018/6510159. eCollection 2018. PMID 30534349
- [Background] Lima AMCT, da Silva Sergio LP, de Souza da Fonseca A. Photobiomodulation via multiple-wavelength radiations. Lasers Med Sci. 2020 Mar;35(2):307-316. doi: 10.1007/s10103-019-02879-1. Epub 2019 Sep 16. PMID 31523781
- [Background] Mosca RC, Ong AA, Albasha O, Bass K, Arany P. Photobiomodulation Therapy for Wound Care: A Potent, Noninvasive, Photoceutical Approach. Adv Skin Wound Care. 2019 Apr;32(4):157-167. doi: 10.1097/01.ASW.0000553600.97572.d2. PMID 30889017
- [Background] Leyane TS, Jere SW, Houreld NN. Cellular Signalling and Photobiomodulation in Chronic Wound Repair. Int J Mol Sci. 2021 Oct 18;22(20):11223. doi: 10.3390/ijms222011223. PMID 34681882
- [Background] de Sousa AP, Paraguassu GM, Silveira NT, de Souza J, Cangussu MC, dos Santos JN, Pinheiro AL. Laser and LED phototherapies on angiogenesis. Lasers Med Sci. 2013 May;28(3):981-7. doi: 10.1007/s10103-012-1187-z. Epub 2012 Aug 25. PMID 22923269
- [Background] Moskvin SV, Geynitz AV, Askhadulin EV. Efficiency of a New Combined Laser Therapy in Patients With Trophic Ulcers of Lower Extremities and Chronic Venous Insufficiency. J Lasers Med Sci. 2017 Summer;8(3):132-135. doi: 10.15171/jlms.2017.24. Epub 2017 Jun 27. PMID 29123633
- [Background] de Lima FJ, Barbosa FT, de Sousa-Rodrigues CF. Use alone or in Combination of Red and Infrared Laser in Skin Wounds. J Lasers Med Sci. 2014 Spring;5(2):51-7. PMID 25653799
- [Background] Santos NR, de M Sobrinho JB, Almeida PF, Ribeiro AA, Cangussu MC, dos Santos JN, Pinheiro AL. Influence of the combination of infrared and red laser light on the healing of cutaneous wounds infected by Staphylococcus aureus. Photomed Laser Surg. 2011 Mar;29(3):177-82. doi: 10.1089/pho.2009.2749. Epub 2011 Jan 8. PMID 21214389